CLINICAL TRIAL: NCT07338318
Title: Effects of E-Cigarette Use on Oxidative and Matrix-Degrading Pathways in Periodontally Healthy Tissues
Brief Title: Effects of E-Cigarette Use on Oxidative Stress and Matrix Degradation
Acronym: ECIG-FOXO
Status: Completed | Type: Observational
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Zeliha Guney, Associate prof., Ankara Medipol University
Other Study IDs: AnkaraMedipolUni.; 16.04.2025/80 (Other: Ankara Medipol University Non-Interventional Clinical Research Ethics Committee)
Record Dates: First submitted 2026-01-03; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-04

CONDITIONS: Smoking Behaviors; Periodontal Health
Keywords: e-cigarette; periodontal health; matrix metalloproteinaz-9; forkhead-box protein 1
MeSH Terms: conditions — Smoking; Vaping | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Gingival crevicular fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- E-Cigarette Users: Participants who have used electronic cigarettes exclusively for at least 12 months, with no history of conventional cigarette use during that period. Eligible individuals must report daily vaping habits and nicotine-containing e-liquid use. All participants will present with clinically healthy periodontal tissues,
  Interventions: Other: E-Cigarette Use

INTERVENTIONS:
Other: E-Cigarette Use — Exclusive e-cigarette users for at least 12 consecutive months, with no conventional cigarette or other tobacco product use during that period. Participants report daily vaping of nicotine-containing e-liquids using refillable or disposable e-cigarette devices. The group represents chronic exposure to aerosolized nicotine and flavoring agents without combustion products

SUMMARY:
This cross-sectional observational study aims to investigate the effects of e-cigarette use on oxidative and matrix-degrading pathways in periodontally healthy individuals. Gingival crevicular fluid biomarkers, including matrix metalloproteinase-9 (MMP-9), reactive oxygen species (ROS), and forkhead-box-1 (FOXO1), will be analyzed to compare the biochemical and inflammatory responses among three groups: e-cigarette users, conventional cigarette smokers, and non-smokers. The study seeks to clarify whether e-cigarette use induces subclinical inflammatory or proteolytic activity in oral tissues comparable to that of traditional smoking.

DETAILED DESCRIPTION:
Cigarette smoking is a well-established risk factor for periodontal tissue destruction, primarily through oxidative stress and upregulation of proteolytic enzymes such as matrix metalloproteinases (MMPs). The advent of electronic cigarettes (e-cigarettes) has introduced an alternative nicotine delivery system, often perceived as less harmful due to the absence of combustion. However, the biological effects of e-cigarette aerosols on oral and periodontal tissues remain unclear.

Matrix metalloproteinase-9 (MMP-9) and reactive oxygen species (ROS) are key enzymes involved in extracellular matrix degradation and the regulation of oxidative stress, respectively. Both biomarkers are found in gingival crevicular fluid (CGF) and are elevated during inflammatory conditions, including periodontitis and peri-implant diseases. Evidence suggests that conventional cigarette smoking increases salivary MMP-9 and ROS levels, reflecting enhanced oxidative and enzymatic tissue breakdown. Whether similar alterations occur in exclusive e-cigarette users with clinically healthy periodontal tissues remains to be determined.

The ECIG study is a cross-sectional, observational clinical investigation designed to evaluate oxidative and matrix-degrading pathways in periodontally healthy individuals across three groups: e-cigarette users, conventional smokers, and non-smokers. GCF samples will be collected to assess biochemical markers, including MMP-9, ROS, and total antioxidant capacity, using ELISA-based methods. Standardized periodontal parameters (plaque index, gingival index, probing depth, and clinical attachment level) will be recorded to confirm periodontal health status.

This study aims to test the hypothesis that exclusive e-cigarette use induces measurable oxidative and proteolytic activity in GCF, comparable to that observed in conventional smokers, despite the absence of clinical periodontal inflammation. Understanding these mechanisms may provide valuable insights into the subclinical impact of vaping on oral health and contribute to public health discussions regarding the relative safety of e-cigarette use.

ELIGIBILITY:
Inclusion Criteria:

* E-cigarette using, conventional smokers, non-smokers

Exclusion Criteria:

* Having active periodontal disease, systemic health problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Systemically and periodontally healthy smokers, e-cigarette users, and non-smoking individuals over 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
(MMP-9, ROS, FOXO-1) Concentration in GCF | Single measurement at baseline (cross-sectional assessment)
  MMP-9, ROS, FOXO-1 levels will be quantified using a commercially available enzyme-linked immunosorbent assay (ELISA) to assess proteolytic activity in periodontally healthy individuals. The mean MMP-9, ROS, and FOXO-1 concentrations (ng/mL) will be compared among three groups: exclusive e-cigarette users, conventional smokers, and non-smokers.

SECONDARY OUTCOMES:
correlation clinical parameters and gcf biomarkers | single time point
  Clinical periodontal indices will be correlated with the expression levels of MMP-9, ROS, and foxo-1.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Medipol Uni., Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. Only summary and aggregated data relevant to the study outcomes will be published in scientific journals or presented at academic meetings. Data sharing beyond this is not planned due to participant confidentiality and ethical restrictions set by the Ankara Medipol University Non-Interventional Clinical Research Ethics Committee